CLINICAL TRIAL: NCT01120080
Title: Advancing Tobacco and Cancer Control: Reducing Alcohol Use to Promote Smoking Cessation
Brief Title: Alcohol Counseling for Telephone Quitline Callers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 091105931; 091105931 (Other: Yale Univ. School of Medicine Human Investigation Committee); R01CA140256 (NIH)
Record Dates: First submitted 2010-04-26; First posted 2010-05-10 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2013-01

CONDITIONS: Smoking; Nicotine Dependence; Alcohol Dependence
Keywords: Smoking; Tobacco; Drinking
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Practical Counseling (Placebo Comparator)
  Interventions: Behavioral: Practical Counseling
- Alcohol Intervention Counseling (Active Comparator)
  Interventions: Behavioral: Alcohol Intervention Counseling

INTERVENTIONS:
Behavioral: Practical Counseling — To ensure that treatment effects are not due to the longer counseling intervention and additional alcohol intervention workbook in the Alcohol Intervention plus Standard Care condition, we will provide additional smoking cessation advice that will not be specific to alcohol use and an additional smoking cessation workbook for participants in the Practical Counseling plus Standard Care condition. Consistent with the Clinical Practice Guideline Update, we will include 5 minutes of practical counseling, which has been shown empirically to be effective in improving rates of smoking cessation.
  Arms: Practical Counseling
Behavioral: Alcohol Intervention Counseling — The Alcohol Intervention counseling protocol will be adapted from Dr. Ockene's brief alcohol intervention protocol and Dr. Kahler's brief alcohol intervention for smokers: Feedback and discussion on the relationship between drinking and smoking, and on the potential effects of alcohol consumption on smoking cessation; an emphasis on personal Responsibility for choosing to change one's behavior; Advice to avoid or minimize drinking during the smoking cessation process; a Menu of options for carrying out a change strategy; use of Empathy by the clinician; and encouragement of Self-efficacy (i.e., confidence) for successful change.
  Arms: Alcohol Intervention Counseling

SUMMARY:
The goal of this study is to train phone counselors working for the New York (NY) State Smokers' Quitline to advise callers who drink at hazardous levels to limit or abstain from alcohol use to determine whether this improves smoking cessation outcomes so that we can establish effect size estimates for a full scale multi-site trial.

DETAILED DESCRIPTION:
This is a developmental study to: 1) create and beta test an alcohol counseling protocol with 25 Quitline callers and 2) train Quitline Specialists to provide an alcohol intervention using at least 100 pilot Quitline callers to ensure that Specialists in the alcohol intervention + standard care condition provide counseling that addresses hazardous drinking with a high level of alcohol intervention strategies and skill. After this phase of the study is complete, a developmental randomized clinical trial will be conducted with 1,948 NY Quitline callers who drink at hazardous levels to compare practical counseling + smoking cessation print materials added to standard care (PC + SC condition) to alcohol intervention counseling + alcohol-focused print materials added to standard care (AI + SC condition). Efficacy data from this trial will be used to determine effect size estimates for both quitdate and 7-month self-reported point prevalence abstinence rates. Reduction in alcohol consumption and reduced drinking as a mediator of smoking cessation outcome will be secondary outcomes. Other mediators and moderators of alcohol intervention effects will also be examined as an exploratory outcome. If the effect size estimates are sufficiently large and medically important to pursue a definitive trial, these data will be used to propose a full scale multi-site large study. If an alcohol intervention is shown to enhance treatment outcome in a large-scale study, alcohol interventions with quitline counselors could be translated for use by the entire NY state quitline and other quitlines across the country. This may increase the effectiveness of quitline interventions and thus has the potential to reach millions of smokers, thereby bolstering tobacco and cancer control efforts across the United States.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18+ years)
* Cigarette smokers requesting assistance with quitting smoking
* Hazardous drinkers (per NIAAA criteria)

Exclusion Criteria:

* Eligible for Enhanced Services Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1948 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of advice to limit or abstain from alcohol use in improving smoking cessation. | 6 Months
  To determine if advice to limit or abstain from alcohol use results in improved smoking cessation outcomes in 1,950 smokers who drink at hazardous levels and are calling a telephone Quitline.

SECONDARY OUTCOMES:
Efficacy of advice to limit or abstain from alcohol use. | 6 Months
  To determine if advice to limit or abstain from alcohol use results in reduced alcohol consumption in 1,950 smokers who drink at hazardous levels and are calling a telephone Quitline.
Does reductions in alcohol use mediate smoking cessation success | 6 Months
  To determine if reduction in alcohol use mediates smoking cessation success in 1,950 smokers who drink at hazardous levels and are calling a telephone Quitline.
What factors that determine smoking cessation success also determine who is more likely to respond to the alcohol intervention | 6 Months
  To examine other mediators and moderators of smoking cessation effects to determine which factors and subgroups are more likely to respond to the alcohol intervention and discern mechanisms of treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin A. Toll, Ph.D., Principal Investigator — Yale University
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Toll BA, Martino S, O'Malley SS, Fucito LM, McKee SA, Kahler CW, Rojewski AM, Mahoney MC, Wu R, Celestino P, Seshadri S, Koutsky J, Hyland A, Cummings KM. A randomized trial for hazardous drinking and smoking cessation for callers to a quitline. J Consult Clin Psychol. 2015 Jun;83(3):445-54. doi: 10.1037/a0038183. Epub 2014 Nov 24. PMID 25419583